CLINICAL TRIAL: NCT03262506
Title: Evaluation of Adherence and Engagement in a Cognitive Training Program for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Chief Investigator, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASASTEL study
Record Dates: First submitted 2017-06-07; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Training (Experimental)
  Interventions: Other: Computerized cognitive training

INTERVENTIONS:
Other: Computerized cognitive training — The cognitive training program consists of a set of computerized exercises designed to improve the speed and accuracy of auditory information processing while engaging neuromodulatory systems involved in attention and reward. These exercises continuously adjust the difficulty level to user performance to maintain an approximately 85% rate of correct responses. Trials with correct responses are rewarded with points and animations.

SUMMARY:
There is evidence that computerized cognitive training can improve cognition in healthy older adults and in people at risk of developing dementia, although an effective model to implement the training in the daily life of people and to ensure engagement is missing. This project studies the adherence, engagement and progress on computerized cognitive training exercises that were offered by the Association of Retirees from the Telecommunications (ASASTEL) to its associates. One hundred subjects in three different cities (Rio de Janeiro, Belo Horizonte and Brasilia) received licenses to perform the exercises on line and were followed by a team of psychologists. We will evaluate adherence, engagement and progress on the computerized cognitive training exercises of those subjects.

ELIGIBILITY:
Inclusion Criteria:

* To be an associate of ASASTEL, or the spouse of an associate,
* To have access to the internet at home and proficiency on accessing and navigating the internet,
* Availability to be evaluated and followed by the professional team.

Exclusion Criteria:

* Any medical condition that precludes performing the computerized training exercises,
* Score below 27 points in the Mini Mental State Examination (MEEM),
* Moderated or advanced dementia.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Training adherence | 1 year
  Training adherence will be defined as a continuous variable (number of hours of training completed by the participant).

SECONDARY OUTCOMES:
Individual gains on the computerized exercises | 1 year
  The computerized cognitive training platform, called BrainHQ, provided by Posit Science Inc, provides the individual gains on the computerized exercises with training.
Motivation with the computerized training exercise | 1 year
  Motivation will be assessed by quantitative (measured as a percentage of all stimulus sets available in the exercises of the BrainHq computerized cognitive training platform) and qualitative questionnaires (Adapted Ultrech Engagement Scale - UWES).
Training adherence (dichotomic variable) | 1 year
  Additionally training adherence will be defined as a dichotomic variable (below or above 10 hours of training).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No